CLINICAL TRIAL: NCT03956524
Title: An Open-label, Comparative, Clinical Phase 1 Study to Assess the Safety and Tolerability of Typhoid Conjugate Vaccine (EuTCV) in Healthy Adults
Brief Title: Safety and Tolerability of Typhoid Conjugate Vaccine (EuTCV) in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EuBiologics Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UTCV_101
Record Dates: First submitted 2019-05-15; First posted 2019-05-20 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Typhoid Fever
MeSH Terms: conditions — Typhoid Fever | interventions — Vi polysaccharide vaccine, typhoid

STUDY DESIGN:
Intervention Model Description: Healthy adult volunteers will be randomized in a 1:1:1 ratio to receive single dose of test or the comparator vaccines.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test group (Experimental): Single dose of EuTCV will be administered intramuscularly
  Interventions: Biological: EuTCV
- Comparator group 1 (Active Comparator): Single dose of Typbar-TCV™ will be administered intramuscularly
  Interventions: Biological: Typbar-TCV™
- Comparator group 2 (Active Comparator): Single dose of Typhim Vi® will be administered intramuscularly
  Interventions: Biological: Typhim Vi®

INTERVENTIONS:
Biological: EuTCV — Single 0.5 mL dose of TCV of EuBiologics co., Ltd.
  Arms: Test group
Biological: Typbar-TCV™ — Single 0.5 mL dose of TCV of Bharat Biotech
  Arms: Comparator group 1
Biological: Typhim Vi® — Single 0.5 mL dose of Vi capsular polysaccharide vaccine of Sanofi Pasteur
  Arms: Comparator group 2

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of EuTCV, in comparison to TCV (Typbar-TCV™, Bharat Biotech) and Vi-Polysaccharide vaccine (Typhim Vi®, Sanofi Pasteur) in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged between and including 18 and 45 years at time of Visit 1
2. Subjects willing to give written informed consent to participate in the trial
3. Subjects who are healthy as determined by medical history, with no clinically significant abnormalities in clinical examination and laboratory tests

Exclusion Criteria:

1. Subjects unwilling to give his/her consent to participate in the trial
2. Subjects who have received Typhoid containing vaccines
3. Subjects who have past history of Typhoid
4. Subjects already immunized with any licensed vaccine within 4 weeks
5. Subjects with known hypersensitivity to any component of the study vaccine
6. Subjects who are pregnant, lactating or childbearing age not using a reliable method of contraception
7. Subjects with any abnormality or chronic disease
8. Subjects with evidence of acute illness within past 7 days requiring systemic antibiotic or antiviral therapy
9. Subjects who have experienced transient thrombocytopenia or neurological complications following an earlier immunization against diphtheria and/or typhoid
10. Subjects who have known history of immune function disorders
11. Subjects who have known history of administration of blood or blood-derived products
12. Subjects who have history of alcohol or substance abuse

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2019-03-16 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Local and systemic solicited adverse events | Day 7
Unsolicited adverse events | up to 6 weeks
Serious adverse events | up to 6 weeks

SECONDARY OUTCOMES:
Proportion of subjects with seroconversion | Baseline to Day 42
  Defined as a 4-fold or more rise in anti-Vi antibody titers

CONTACTS AND LOCATIONS:
Locations (1):
- De La Salle Health Sciences Institute, Dasmariñas, Cavite, Philippines

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choi SK, Baik YO, Kim CW, Kim SK, Oh IN, Yoon H, Yu D, Lee C. An open-label, comparative, single dose, clinical Phase Ⅰ study to assess the safety and immunogenicity of typhoid conjugate vaccine (Vi-CRM197) in healthy Filipino adults. Vaccine. 2021 May 6;39(19):2620-2627. doi: 10.1016/j.vaccine.2021.03.089. Epub 2021 Apr 10. PMID 33849723